CLINICAL TRIAL: NCT00108355
Title: Vasoconstrictors as Alternatives to Albumin After Large Volume Paracentesis in Cirrhosis
Brief Title: Vasoconstrictors as Alternatives to Albumin After Large-Volume Paracentesis (LVP) in Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-016-03F; NCT00530959 (obsolete NCT alias)
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-02

CONDITIONS: Ascites; Cirrhosis
Keywords: albumin; ascites; paracentesis
MeSH Terms: conditions — Ascites; Fibrosis | interventions — Albumins; Midodrine; Tablets; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albumin (Control group) (Active Comparator): After LVP, patients in this group received:
  Intravenous albumin (25%) at 8 g/liter of ascitic fluid removed, one time dose; Intramuscular injection of 5 cc saline (Octreotide LAR placebo), every 30 days ; Oral tablet 3 times a day (Midodrine placebo)
  Interventions: Drug: Albumin; Drug: Oral tablet (Midodrine placebo); Drug: Saline injection (Octreotide LAR placebo); Procedure: Large Volume Paracentesis
- Vasoconstrictor (Study Group) (Experimental): After LVP, patients in this group received:
  Octreotide LAR intramuscular injection 20 mg, every 30 days; Midodrine tablet, 10 mg three times a day; Intravenous saline infusion (Albumin placebo), one time dose
  Interventions: Drug: Intravenous Saline Infusion (Albumin placebo); Drug: Midodrine; Drug: Octreotide LAR; Procedure: Large Volume Paracentesis

INTERVENTIONS:
Drug: Albumin — Intravenous Albumin at a dose of 8g/liter of ascitic fluid removed
  Arms: Albumin (Control group)
Drug: Intravenous Saline Infusion (Albumin placebo) — Intravenous saline Infusion (Albumin placebo)
  Arms: Vasoconstrictor (Study Group)
Drug: Midodrine — Midodrine oral tablet at 10 mg three times a day.
  Arms: Vasoconstrictor (Study Group)
Drug: Oral tablet (Midodrine placebo) — Oral tablet (Midodrine placebo) three times a day
  Arms: Albumin (Control group)
Drug: Octreotide LAR — Octreotide LAR 20 mg intramuscular injection every 30 days
  Arms: Vasoconstrictor (Study Group)
Drug: Saline injection (Octreotide LAR placebo) — Saline intramuscular injection 5 cc every 30 days.
  Arms: Albumin (Control group)
Procedure: Large Volume Paracentesis — Procedure to remove large amounts (more than 5 liter) of ascitic fluid via a catheter.
  Other Names: LVP

SUMMARY:
This clinical trial compares a combination of two drugs that constrict blood vessels (Octreotide LAR and Midodrine) to albumin after large volume paracentesis. Subjects have cirrhosis and ascites.

DETAILED DESCRIPTION:
This prospective, placebo-controlled, randomized, clinical trial compares the effect of a combination of vasoconstrictors (octreotide plus midodrine) to albumin on the time to recurrence of ascites in patients with refractory ascites treated with large volume paracentesis. The treatment allocation ratio for the two treatment arms is 1:1 using a stratified random permuted block design. Subjects are patients 18-80 years old with cirrhosis and ascites who are stratified according to the presence or absence of renal dysfunction at the time of randomization. Measurements include blood pressure, weight, girth, abdominal ultrasound, forearm blood flow, plasma renin activity, angiotensin, and aldosterone, repeated during a 6 month period.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of any etiology
* Age 18-80 years
* Moderate to severe ascites

Exclusion Criteria:

* No or small ascites
* Severe hepatic hydrothorax
* Recent GI (gastrointestinal) hemorrhage
* Active bacterial infection
* Cardiac failure
* Organic renal disease
* Hepatocellular carcinoma
* Severe comorbidity (advanced neoplasia)
* Serum creatinine > 3 mg/dl
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2003-12; Primary Completion 2010-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Garcia-Tsao, MD, Principal Investigator — VA Connecticut Health Care System (West Haven)
Locations (1):
- VA Connecticut Health Care System (West Haven), West Haven, Connecticut, United States

REFERENCES:
- [Background] Karwa R, Woodis CB. Midodrine and octreotide in treatment of cirrhosis-related hemodynamic complications. Ann Pharmacother. 2009 Apr;43(4):692-9. doi: 10.1345/aph.1L373. Epub 2009 Mar 18. PMID 19299324
- [Result] Bernardi M, Caraceni P, Navickis RJ, Wilkes MM. Albumin infusion in patients undergoing large-volume paracentesis: a meta-analysis of randomized trials. Hepatology. 2012 Apr;55(4):1172-81. doi: 10.1002/hep.24786. PMID 22095893
- [Result] Moreau R, Asselah T, Condat B, de Kerguenec C, Pessione F, Bernard B, Poynard T, Binn M, Grange JD, Valla D, Lebrec D. Comparison of the effect of terlipressin and albumin on arterial blood volume in patients with cirrhosis and tense ascites treated by paracentesis: a randomised pilot study. Gut. 2002 Jan;50(1):90-4. doi: 10.1136/gut.50.1.90. PMID 11772973
- [Result] Lata J, Marecek Z, Fejfar T, Zdenek P, Bruha R, Safka V, Hulek P, Hejda V, Dolina J, Stehlik J, Tozzi I. The efficacy of terlipressin in comparison with albumin in the prevention of circulatory changes after the paracentesis of tense ascites--a randomized multicentric study. Hepatogastroenterology. 2007 Oct-Nov;54(79):1930-3. PMID 18251131
- [Result] Angeli P, Volpin R, Gerunda G, Craighero R, Roner P, Merenda R, Amodio P, Sticca A, Caregaro L, Maffei-Faccioli A, Gatta A. Reversal of type 1 hepatorenal syndrome with the administration of midodrine and octreotide. Hepatology. 1999 Jun;29(6):1690-7. doi: 10.1002/hep.510290629. PMID 10347109
- [Result] Bari K, Minano C, Shea M, Inayat IB, Hashem HJ, Gilles H, Heuman D, Garcia-Tsao G. The combination of octreotide and midodrine is not superior to albumin in preventing recurrence of ascites after large-volume paracentesis. Clin Gastroenterol Hepatol. 2012 Oct;10(10):1169-75. doi: 10.1016/j.cgh.2012.06.027. Epub 2012 Jul 16. PMID 22801062
- [Result] Appenrodt B, Wolf A, Grunhage F, Trebicka J, Schepke M, Rabe C, Lammert F, Sauerbruch T, Heller J. Prevention of paracentesis-induced circulatory dysfunction: midodrine vs albumin. A randomized pilot study. Liver Int. 2008 Aug;28(7):1019-25. doi: 10.1111/j.1478-3231.2008.01734.x. Epub 2008 Apr 11. PMID 18410283
- [Result] Singh V, Dheerendra PC, Singh B, Nain CK, Chawla D, Sharma N, Bhalla A, Mahi SK. Midodrine versus albumin in the prevention of paracentesis-induced circulatory dysfunction in cirrhotics: a randomized pilot study. Am J Gastroenterol. 2008 Jun;103(6):1399-405. doi: 10.1111/j.1572-0241.2008.01787.x. PMID 18547224
- [Result] Tandon P, Tsuyuki RT, Mitchell L, Hoskinson M, Ma MM, Wong WW, Mason AL, Gutfreund K, Bain VG. The effect of 1 month of therapy with midodrine, octreotide-LAR and albumin in refractory ascites: a pilot study. Liver Int. 2009 Feb;29(2):169-74. doi: 10.1111/j.1478-3231.2008.01778.x. Epub 2008 May 19. PMID 18492024
- [Result] Singh V, Kumar R, Nain CK, Singh B, Sharma AK. Terlipressin versus albumin in paracentesis-induced circulatory dysfunction in cirrhosis: a randomized study. J Gastroenterol Hepatol. 2006 Jan;21(1 Pt 2):303-7. doi: 10.1111/j.1440-1746.2006.04182.x. PMID 16460491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2003 and June 2010, about 200 patients with cirrhosis and ascites were screened, of which, only 29 met inclusion criteria. Twenty five patients (13 control, 12 study group) were included in the analysis.
Groups:
- Vasoconstrictors (Study Group): After LVP, patients in this group received:
  Octreotide LAR intramuscular injection 20 mg, every 30 days; Midodrine tablet, 10 mg three times a day; Intravenous saline infusion (Albumin placebo), one time dose
Period: Overall Study
Arm/Group | Albumin (Control Group) | Vasoconstrictors (Study Group)
Started | 15 (Two patients met inclusion criteria not randomized, one had peritonitis , other loculated ascites.) | 14 (Two patients met inclusion criteria not randomized, one had peritonitis, other loculated ascites.)
Completed | 13 | 12
Not Completed | 2 | 2
Not completed — Peritonitis at index paracentesis | 1 | 1
Not completed — Loculated ascites, limiting paracentesis | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Vasoconstrictor (Treatment Group): After LVP, patients in this group received:
  Octreotide LAR intramuscular injection 20 mg, every 30 days; Midodrine tablet, 10 mg three times a day; Intravenous saline infusion (Albumin placebo), one time dose
- Total: Total of all reporting groups
Arm/Group | Albumin (Control Group) | Vasoconstrictor (Treatment Group) | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 2 | 2 | 4
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  age median | 55 (7.5) [51 to 61] | 60 (8.4) [51 to 65] | 58 (8) [51 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence of Ascites.
Description: Comparison between Albumin (Control group) and Vasoconstrictor (Treatment group)
Time Frame: Variable depending on the patient, average 10 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Albumin (Control Group) | Vasoconstrictor (Treatment Group)
Number analyzed (Participants) | 13 | 12
days | 10 [7 to 29] | 8 [6 to 22]
Statistical Analysis 1: Comparison: Albumin (Control Group) vs Vasoconstrictor (Treatment Group); Initial estimation: median time to recurrence of ascites of 38 days in the study group and 20 days in the control group in a fixed duration of 6 months (5% type-I error (2 sided) and an 80% power). However, due to low accrual and based on randomized trials using vasoconstrictors in the prevention of PCD and a study that showed that midodrine leads to a significant improvement in effective arterial blood volume, each of which had sample sizes of 24-25 patients,we decided on a sample size of 30; Test type: Superiority or Other; p < 0.05, Log Rank

2. Secondary Outcome: Development of Post-paracentesis Circulatory Dysfunction (PCD)
Description: Defined as an increase in Plasma Renin Activity (PRA) by >50% from baseline to a level > 4 ng/mL/h at post-paracentesis day
Time Frame: 6 days after paracentesis
Population: Plasma Renin Activity (lab value to measure PCD) was not available for 6 patients leaving 11 patients in Albumin (control group) and 8 patients in Vasoconstrictor (Treatment group) for this outcome analysis.
Measure: Number; unit: participants
Arm/Group | Albumin (Control Group) | Vasoconstrictor (Treatment Group)
Number analyzed (Participants) | 11 | 8
participants | 2 | 2

ADVERSE EVENTS:
Arm/Group | Albumin (Control Group) | Vasoconstrictor (Treatment Group)
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 3/13 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albumin (Control Group) (N=13) | Vasoconstrictor (Treatment Group) (N=12)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
GI Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Scrotal edema (Renal and urinary disorders) | 1 (1) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Difficulty to enroll patient population lead to small sample size. Midodrine not titrated for a goal increase in mean arterial pressure. Blood tests for day 6 assessment of post paracentesis circulatory dysfunction not available for all patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No